CLINICAL TRIAL: NCT07327333
Title: The Effects of Contextual-Based Augmented Reality Facilitated Education in Promoting Oral Mucositis Care Among Nurses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24MMHIS312e
Record Dates: First submitted 2025-04-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-02

CONDITIONS: Nursing Education
Keywords: Augmented Reality; Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Situational Augmented Reality-Assisted Teaching (Experimental): Using situational augmented reality-assisted teaching as a case, different grades of oral mucositis are presented for learners to perform care for various stages of oral mucositis. Through clinical reasoning, learners select appropriate interventions and directly observe changes and outcomes in the patient's oral mucosa.
  Interventions: Other: Situational Augmented Reality-Assisted Teaching
- Classroom Teaching (Placebo Comparator): Here is the translation in English: "Explain the causes and effects of oral mucositis. Explain the timing of oral mucositis assessment, assessment tools, and how to use them. Explain the different stages of oral mucositis and how to provide appropriate treatment and care for each stage. Share clinical case examples, guide learners to describe the case situations, and encourage them to understand and reflect on how to perform proper assessment and care, and provide feedback to the learners." Explain the causes and effects of oral mucositis. Describe the appropriate timing for oral mucositis assessment, introduce assessment tools, and demonstrate how to use them.
  Discuss the different grades of oral mucositis and how to provide proper treatment and care based on its severity.
  Share real-life clinical cases to guide learners in describing the scenario, understanding and reflecting on how to conduct proper assessment and care, and provide feedback to the learners.
  Interventions: Other: Classroom Teaching

INTERVENTIONS:
Other: Situational Augmented Reality-Assisted Teaching — Using situational augmented reality-assisted teaching as a case study, learners are presented with varying grades of oral mucositis. Learners then perform appropriate care for each grade of mucositis. Through clinical reasoning, they select suitable interventions, and finally, directly observe changes and outcomes in the patient's oral mucosa.
  Arms: Situational Augmented Reality-Assisted Teaching
Other: Classroom Teaching — Classroom Teaching and Case Sharing Introduction to Updated Oral Mucositis Guidelines and Care Management of Common Oral Mucositis Complications Case Sharing on Oral Mucositis Complication Management: Researchers
  Arms: Classroom Teaching

SUMMARY:
In recent years, cancer has become one of the leading causes of death worldwide, with an increasing number of people being diagnosed with the disease. Current cancer treatments include surgery, chemotherapy (CT), radiotherapy (RT), concurrent chemoradiotherapy (CCRT), targeted therapy, immunotherapy, and hematopoietic stem cell transplantation (HSCT). While these treatments have improved survival rates for many patients, they often lead to adverse side effects, one of the most common being oral mucositis (OM). Oral mucositis in cancer patients differs from general types of oral ulcers, primarily caused by the toxicity of chemotherapy drugs and radiation therapy, leading to extensive damage to epithelial cells. This study aims to validate the effectiveness of "situational augmented reality-assisted instruction" in an educational intervention program for oral mucositis care in enhancing nursing personnel's knowledge of oral mucositis care, oral mucositis care abilities, clinical reasoning skills, and learning engagement. A randomized clinical trial (RCT) was conducted using convenience sampling, targeting nursing personnel from cancer-related units at a teaching hospital in northern Taiwan. A follow-up study with repeated measures in two groups was performed. Self-developed scales based on relevant literature and expert recommendations were used to assess knowledge of oral mucositis care and self-evaluated oral mucositis care abilities. Additionally, the Clinical Reasoning Scale (CRS) by Huang et al. (2023) and the Learning Engagement Scale revised by Chiu (2020) were employed as research tools. Data were analyzed using SPSS version 29.0, with descriptive statistics including frequency distribution, percentage, mean, and standard deviation. The results of this study will provide relevant institutions and educational training units with references for the content and assessment of oral mucositis care courses for cancer nursing personnel, and further applications of the research findings.

ELIGIBILITY:
Inclusion Criteria:

* Cancer-related nursing staff from a medical center in northern Taiwan.
* Individuals willing to participate in this study and who have signed the informed consent form.

Exclusion Criteria:

* Nursing staff from non-cancer-related departments or departments not included in the eligibility criteria.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
The Effects of Contextual-Based Augmented Reality Facilitated Education in Promoting Oral Mucositis Care among Nurses | 2 months
  First Outcome Measures: **Oral Mucositis Care Knowledge Scale** This study will assess Oral Mucositis care knowledge using the **Oral Mucositis Care Knowledge Scale**. The scale ranges from **0 to 100**, with higher scores indicating **better** knowledge levels. The assessment will be conducted at **baseline and post-intervention** to measure changes in Oral Mucositis care knowledge over time. Time Frame: 2months.

SECONDARY OUTCOMES:
Clinical Reasoning Scale Description | The scale ranges from 16 to 80, with higher scores representing better clinical reasoning ability. Measurements will be taken before and after the intervention to assess changes in clinical reasoning performance. Time Frame: 6months.

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan